CLINICAL TRIAL: NCT04495400
Title: Percutaneous Screw Fixation vs. Open Fixation in the Treatment of Thoracolumbar Fractures
Acronym: PrecScrew
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Salah Aoun, Assistant Professor, University of Texas Southwestern Medical Center
Other Study IDs: STU 042018-004
Record Dates: First submitted 2020-03-31; First posted 2020-07-31 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Lumbar Vertebral Fracture
MeSH Terms: conditions — Spinal Fractures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Percutaneous Screw Fixation: Patients who have had a Percutaneous Screw fixation procedure.
  Interventions: Procedure: Thoracolumbar Fracture Fixation
- Open Fixation: Patients who have had an Open Fixation procedure.
  Interventions: Procedure: Thoracolumbar Fracture Fixation

INTERVENTIONS:
Procedure: Thoracolumbar Fracture Fixation — The is surgery is preformed on patients who have had a blunt trauma fractures between the T10 and the L2. The surgical management for more severe/unstable fractures usually involves posterior instrumentation with percutaneous or open pedicle screw fixation. While the traditional open pedicle screw fixation technique has demonstrated good radiologic and clinical outcomes, a minimally invasive percutaneous approach has been increasingly used in recent years.

SUMMARY:
In this single-center retrospective study, the investigators will include all patients admitted to Parkland Hospital who underwent surgical fixation of thoracolumbar fractures between the years 2000 and 2017. The study investigators will gather demographic, radiographic, and operative information. Patients will be matched according to demographic information in a case-control style. The primary outcome of the study will be comparing the clinical and radiographic outcomes of two surgical techniques in order to establish the best treatment approach for this disease.

DETAILED DESCRIPTION:
Thoracolumbar (TL) fractures occur in 8-15% of blunt trauma patients cared for in major trauma centers. These fractures can be devastating and commonly occur in patients who endure high-energy trauma (e.g. motor vehicle accidents). TL fractures occur mainly between T10 and L2. The "3 Column Model" attempts to identify criteria that can predict instability of TL fractures. This model divides the spine into anterior, middle, and posterior areas. Stability is dependent on the integrity of two out of three of the columns. Major spine injuries are those that involve mechanical or neurologic instability.

The four major types of injury include compression, burst, seat-belt, and fracture-dislocation. Compression fractures account for 50-70% of all TL fractures and usually consist of compression failure of the anterior column. Burst fractures comprise approximately 14% of all TL injuries. These injuries usually involve compression of both the anterior and posterior column. Seat-belt fractures (aka flexion-distraction fractures) account for 10% of TL injuries and occur most commonly in patients who are wearing only the lap belt (i.e. no chest belt) during motor vehicle trauma. These injuries typically involve compression of the anterior column with distraction failure of both the middle and posterior columns. Finally, the fracture-dislocation type fracture occurs with massive direct trauma to the back, causing failure of all three columns and translational injury.

Patients with TL fractures may present with TL spine pain, midline TL spine tenderness, TL spine bony deformity, or neurologic deficit. Oftentimes these patients were in high-velocity traumatic scenarios, including falls from heights, crush injuries, motor vehicle crashes with ejection, unenclosed vehicles (ex. motorcycles), or automobile versus pedestrian accidents. Diagnosis is confirmed via computed tomography (CT) imaging or plain radiographs. CT imaging is typically more accurate than plain radiographs but can be poor in certain subtypes of injury. MRI can be utilized to assess the integrity of the ligaments and surrounding soft tissues.

There is currently no universally accepted system for classifying the severity of TL fractures. One proposed system is the Thoracolumbar injury classification and severity score (TLICS). Points are awarded based on radiographic findings, neurologic status, and the integrity of posterior ligamentous complex. The final numeric score is used to guide treatment, with higher scores indicating need for surgery. Neurologic deficit favors surgery.

There is no clear consensus on the best treatment approach for TL fractures. For situations where conservative management is decided (i.e. surgery is not required or is contraindicated), patients are treated with recumbency and delayed ambulation in orthosis with serial radiographs to determine need for further intervention. The surgical management for more severe/unstable fractures usually involves posterior instrumentation with percutaneous or open pedicle screw fixation.3 While the traditional open pedicle screw fixation technique has demonstrated good radiologic and clinical outcomes, a minimally invasive percutaneous approach has been increasingly used in recent years. The minimally invasive technique potentially carries the advantage of less operative blood loss, shorter operative time, smaller incisions, potentially less postoperative pain, and overall shorter hospital stay. There are a few studies published in the literature, but more studies are needed to establish the treatment modality that is the most efficacious and safe for these patients.

At the University of Texas Southwestern (Parkland Hospital), the investigators evaluate and treat a large population of patients with TL fractures. Previous trials in the literature comparing open and percutaneous fixation of TL fractures have been series of ~100-200 patients. These studies have shown variable results, with many concluding similar outcome results for the two surgical techniques. The purpose of this study is to compare a larger number of patients (~500) who have undergone either surgical approach to determine the best technique in terms of clinical and radiographic outcomes. The investigators believe this study will provide neurosurgeons with invaluable information about the safety and efficacy of different treatment modalities for TL fractures in this patient population.

ELIGIBILITY:
Inclusion Criteria:

Patients with thoracolumbar fractures:

* Who underwent open surgical fixation at Parkland Hospital
* Who underwent percutaneous (minimally invasive) screw fixation at Parkland Hospital • Age above 18 years

Exclusion Criteria:

* Age below 18
* Bleeding disorders
* Prior surgical fixation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients from 200 to 2017 who have either had a Percutaneous fixation or an open fixation for thoracolumbar fractures
Sampling Method: Non-Probability Sample
Enrollment: 485 (Actual)
Dates: Start 2018-04-23 (Actual); Primary Completion 2019-09-19 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Rate of Positive and Negative Clinical Outcomes based on hospital adverse events | 2000-2017
  Hospital Adverse Events
Rate of positive and negative radiographic outcomes based on cobb angle of kyphosis and vertebral wedge angle | 2000-2017
  Curvature of spine post-surgery

CONTACTS AND LOCATIONS:
Overall Officials: Salah Aoun, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Parkland Health and Hospital System, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared.